CLINICAL TRIAL: NCT01623258
Title: A Prospective Randomized Study Comparing Sentinel Lymph Node (SLN) Evaluation With Standard Pathological Evaluation for the Staging of Colon Carcinoma
Status: Completed | Type: Observational
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alexander Stojadinovic, Chief, Surgical Oncology, Walter Reed Army Medical Center
Other Study IDs: 03-20010
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard of Care: Standard histopathological evaluation using conventional paraffin embedding, sectioning and hematoxylin and eosin staining and microscopy without sentinel lymph node ultrastaging
- Research: SOC with sentinel lymph node analysis

SUMMARY:
The objective of this trial is to define the rate of upstaging of colon carcinoma lymph node metastasis with sentinel lymph node (SLN) mapping.

Null hypothesis: There is no difference in the rate of lymph node metastasis between conventional histopathological processing of lymph nodes and SLN mapping with detailed pathologic examination using immunohistochemistry (IHC) in patients undergoing resection of colon carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age
2. Primary, non-metastatic [Stage I, II (localized, node negative), or III (localized, node positive)] colon carcinoma confirmed by tissue biopsy or colon mass clinically consistent with cancer and eventually confirmed by pathology
3. Palpable mass at time of surgery
4. Capable of providing informed consent

Exclusion Criteria:

1. Prior radiation or chemotherapy
2. Non-palpable colon tumor
3. Recurrent or Stage IV (metastatic) colon cancer
4. Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 150 male or female military healthcare beneficiaries over the age of 18 years presenting at the Walter Reed Army Medical Center (WRAMC) General Surgery clinic with the diagnosis of biopsy-proven, primary, non-metastatic (Clinical Stage I,II or III) colon carcinoma will be enrolled. Subjects with colonic masses clinically consistent with colon cancer, and eventually confirmed by pathology, will also be enrolled.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2002-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Define the rate of upstaging of colon carcinoma lymph node metastasis with define the rate of upstaging of colon carcinoma lymph node metastasis with sentinel lymph node (SLN) mapping | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stojadinovic, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Nissan A, Protic M, Bilchik AJ, Howard RS, Peoples GE, Stojadinovic A. United States Military Cancer Institute Clinical Trials Group (USMCI GI-01) randomized controlled trial comparing targeted nodal assessment and ultrastaging with standard pathological evaluation for colon cancer. Ann Surg. 2012 Sep;256(3):412-27. doi: 10.1097/SLA.0b013e31826571c8. PMID 22871988